CLINICAL TRIAL: NCT06253741
Title: "Comparison of Rhomboid Intercostal and Subserratus Plane Blocks Applied for Postoperative Analgesia in Video-Assisted Thoracoscopic Surgery With Thoracic Paravertebral Block"
Brief Title: Rhomboid Intercostal and Subserratus / Paravertebral Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Seda Cansabuncu, Medical Doctor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2022-17/23
Record Dates: First submitted 2024-02-01; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Analgesia; Thoracic; Anesthesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PARAVERTEBRAL BLOCK (Active Comparator): After induction of general anesthesia and endotracheal intubation in the operating room, following the positioning of the patient for surgery, ultrasound-guided paravertebral block (PVB) will be routinely performed in our clinic using 0.25% bupivacaine solution at a dose of 0.5 ml/kg.
  Interventions: Procedure: PARAVERTEBRAL BLOCK
- RHOMBOID INTERCOSTAL AND SUBSERRATUS PLANE BLOCK (Active Comparator): After induction of general anesthesia and endotracheal intubation in the operating room, following the positioning of the patient for surgery, rhomboid intercostal block with sub-serratus plane block (RISS) will be routinely performed in our clinic using 0.25% bupivacaine solution at a dose of 0.5 ml/kg under ultrasound guidance.
  Interventions: Procedure: RHOMBOID INTERCOSTAL AND SUBSERRATUS PLANE BLOCK
- PLACEBO (Placebo Comparator): The group without any peripheral block application will be included
  Interventions: Procedure: PLACEBO

INTERVENTIONS:
Procedure: PARAVERTEBRAL BLOCK — Hemodynamic data (mean arterial pressure, heart rate, oxygen saturation) will be recorded for all patients every 30 minutes during the intraoperative period, along with the amount of opioids used throughout the surgery. A patient-controlled analgesia device (PCA) will be connected to each patient 15 minutes before awakening, prepared with a 1mg/ml morphine solution, with a bolus dose of 2 ml and a lockout period of 15 minutes
  Other Names: PVB
  Arms: PARAVERTEBRAL BLOCK
Procedure: RHOMBOID INTERCOSTAL AND SUBSERRATUS PLANE BLOCK — Hemodynamic data (mean arterial pressure, heart rate, oxygen saturation) will be recorded for all patients every 30 minutes during the intraoperative period, along with the amount of opioids used throughout the surgery. A patient-controlled analgesia device (PCA) will be connected to each patient 15 minutes before awakening, prepared with a 1mg/ml morphine solution, with a bolus dose of 2 ml and a lockout period of 15 minutes.
  Other Names: RISS
  Arms: RHOMBOID INTERCOSTAL AND SUBSERRATUS PLANE BLOCK
Procedure: PLACEBO — Hemodynamic data (mean arterial pressure, heart rate, oxygen saturation) will be recorded for all patients every 30 minutes during the intraoperative period, along with the amount of opioids used throughout the surgery. A patient-controlled analgesia device (PCA) will be connected to each patient 15 minutes before awakening, prepared with a 1mg/ml morphine solution, with a bolus dose of 2 ml and a lockout period of 15 minutes.
  Other Names: PG
  Arms: PLACEBO

SUMMARY:
Postoperative pain is a significant concern following video-assisted thoracoscopic surgery (VATS). Pain after thoracic surgery not only causes a strong stress reaction and adverse emotional experience but also affects postoperative rehabilitation. Hence, different analgesia techniques, including local anesthetic infiltration, intercostal nerve block, paravertebral block, and thoracic epidural anesthesia, have been described to attenuate the intensity of acute postoperative painparavertebral block (PVB) and Rhomboid intercostal block with sub-serratus plane block (RISS) are the two types of plane blocks used for postoperative analgesia after video-assisted thoracoscopic surgery (VATS). This prospective randomized controlled trial was performed to analyze the postoperative analgesic effects of ultra- sound-guided PVB and RISS block after video-assisted thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Planned for VATS
* American Society of Anesthesiologists (ASA) class I and II
* Patients aged between 18-80

Exclusion Criteria:

* Contraindications to local anesthetic allergy or bupivacaine
* Known or suspected coagulopathy
* Injection site infection
* History of thoracic surgery
* Severe neurological or psychiatric disorder
* Severe cardiovascular disease
* Liver failure
* Renal failure (glomerular filtration rate <15 ml/min/1.73 m2)
* Chronic opioid use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
VAS scores | up to 24 hours
  The primary outcome of this study was to compare the analgesia of paravertebral block versus rhomboid intercostal and subserratus plane block in VATS surgery.

SECONDARY OUTCOMES:
morphine consumption | up to 24 hours
  The secondary outcome measure in this study was 24-hour morphine consumption.
first analgesia requirement | up to 24 hours
  Secondary outcome measures included time to first request for morphine
Side effects | up to 24 hours
  Side effects associated with morphine consumption

CONTACTS AND LOCATIONS:
Overall Officials: SEDA CANSABUNCU, Principal Investigator — Uludag University
Locations (1):
- Bursa Uludag University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No